CLINICAL TRIAL: NCT06408077
Title: Regulation of Extracellular Sodium in End Stage Renal Disease Upon Volume and Electrolyte Challenges - a Prospective Trial.
Brief Title: Regulation of Extracellular Sodium in End Stage Renal Disease Upon Volume and Electrolyte Challenges
Acronym: RESERVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Volker Burst, Prof. Dr. med., University of Cologne
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: V1.2_2023-06-06
Record Dates: First submitted 2024-05-03; First posted 2024-05-09 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hyponatremia
Keywords: hyponatremia; prospective trial; intracellular measurements; Water-Electrolyte Imbalance
MeSH Terms: conditions — Hyponatremia; Water-Electrolyte Imbalance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Water-Group (Experimental): Intravenous administration of water (Aqua ad injectabilia) until a decrease of plasma sodium of 5 to 8 mmol/l has been achieved
  Interventions: Other: Water administration
- NaCl-Group (Experimental): Intravenous administration of NaCl 3% until an increase of plasma sodium of 5 to 8 mmol/l has been achieved
  Interventions: Other: NaCl-Administration

INTERVENTIONS:
Other: Water administration — Intravenous administration of water (Aqua ad injectabilia) until a decrease of plasma sodium of 5 to 8 mmol/l has been achieved
  Arms: Water-Group
Other: NaCl-Administration — Intravenous administration of NaCl 3% until an increase of plasma sodium of 5 to 8 mmol/l has been achieved
  Arms: NaCl-Group

SUMMARY:
Hyponatremia is the most common electrolyte disorder of all and can be observed in more than 30% of all patients in hospitals. Osmotic homeostasis of body fluids is essential for survival of all living creatures. It is widely accepted that extra- and intracellular osmolalities are in equilibrium at all times and thus, changes in the extracellular osmolality will lead to either shrinkage or swelling of cells which can be detrimental. In severe cases, it can lead to swelling of the brain and death. Even in less dramatic scenarios, symptoms such as epileptic seizures, headaches, depression and dizziness exist, leading to an increased risk of fractures, hospital admissions and a considerable burden for affected patients.

As short-term defense against osmotic stress, each individual cell is capable of actively externalizing or internalizing osmotically active solutes which restores normal or near-normal cell volume at the expense of an altered milieu interior. Obviously, there must be limitations to this strategy if intracellular integrity is meant to be kept stable. It has therefore been postulated that, apart from this cell-immanent mechanism, extracellular and intracellular electrolyte stores could assist in buffering osmotic imbalances.

The Edelman formula states that extracellular sodium is determined by the total amount of exchangeable body sodium (the major extracellular cation) plus potassium (the major intracellular cation) divided by total body water. Several studies have shown, that it only partially explains the changes in patients outside the osmotic equilibrium.

To better understand these physiological responses might not only promote the researcher's insight into the most basic cellular self-defense systems by measuring and comparing extra- and intracellular electrolyte concentrations with estimated changes in a patient that will be intravenously challenged with either water or sodium chloride 3%.

The evolution over time of extra- and intracellular sodium and other electrolytes will be assessed quantitatively in patients with impaired renal function after water or sodium chloride (NaCl) administration.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years
* Requirement of renal replacement therapy due to surgical (i.e., nephrectomy) or non-surgical (chronic kidney disease) reason
* Stable hemodialysis treatment for at least 3 months
* Urine output <100ml in 24 hours
* Glucose-corrected plasma sodium between 135 mmol/l and 145 mmol/l
* Plasma potassium between 3.5 mmol/l and 5 mmol/l
* Written informed consent

Exclusion Criteria:

* Peritoneal dialysis patients
* Signs of volume expansion or contraction
* Congestive heart failure (NYHA ≥2)
* acute illness (infection, congestive heart failure, liver cirrhosis, etc.) requiring hospital admission
* Uncontrolled arterial hypertension
* Hemoglobin ≤8g/dL
* Alcohol abuse
* Malnutrition
* Persons, who are in a dependency/employment relationship with the investigators
* Accommodation in an institution by judicial or administrative order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
acute changes of extracellular osmolality | 300 minutes after infusion
  The primary aim is to compare the actual acute change of extracellular sodium with the estimated change of extracellular sodium in response to an intravenous challenge with either water or sodium. Precise evaluation of the validity of the concept of Edelman in acute changes of extracellular osmolality

SECONDARY OUTCOMES:
change of extracellular electrolyte concentrations | 300 minutes after infusion
  extracellular electrolyte concentrations in response to an intravenous challenge with either water or sodium.
change of intracellular electrolyte concentrations | 300 minutes after infusion
  intracellular (red blood cells/white blood cells) electrolyte concentrations in response to an intravenous challenge with either water or sodium.
change of osmolality | 300 minutes after infusion
  change of osmolality in response to an intravenous challenge with either water or sodium
change of cell volume | 300 minutes after infusion
  cell volume (red blood cells) in response to an intravenous challenge with either water or sodium

CONTACTS AND LOCATIONS:
Overall Officials: Volker Burst, MD, Principal Investigator — University Hospital of Cologne
Locations (1):
- Department II of Internal Medicine,University of Cologne, Cologne, Germany